CLINICAL TRIAL: NCT04749108
Title: Multicentric Phase II-III Study Evaluating the Tailored Management of Locally-advanced Rectal Carcinoma After a Favorable Response to Induction Chemotherapy
Brief Title: Study Evaluating the Tailored Management of Locally-advanced Rectal Carcinoma
Acronym: GRECCAR14
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROICM 2021-01 GRE; 2021-000414-41 (EudraCT Number)
Record Dates: First submitted 2021-02-05; First posted 2021-02-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Locally Advanced Malignant Neoplasm; Rectal Carcinoma
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Drug: Induction chemotherapy - modified FOLFIRINOX regimen Other: Early tumor response evaluation by MRI volumetry Radiation: Radiochemotherapy Cap 50 Procedure: Radical proctectomy with total mesorectal excision
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Arm A: immediate rectal surgery (Experimental): "Very good" responder patients will be randomly assigned to proctectomy performed within 4 to 6 weeks from randomization.
  Interventions: Drug: Induction chemotherapy - modified FOLFIRINOX regimen; Other: Early tumor response evaluation by MRI volumetry; Procedure: Radical proctectomy with total mesorectal excision
- RCT Cap 50 and then rectal surgery (Active Comparator): Very good" responder patients will be randomly assigned to receive chemoradiotherapy combining the administration of oral capecitabine (1600 mg/m2/day, BID) and radiotherapy at a total dose of 50 grays (2Gy/day, 5 days a week, 5 weeks, boost 6 Gy) followed after 7 weeks by a proctectomy.
  Interventions: Drug: Induction chemotherapy - modified FOLFIRINOX regimen; Other: Early tumor response evaluation by MRI volumetry; Radiation: Radiochemotherapy Cap 50; Procedure: Radical proctectomy with total mesorectal excision

INTERVENTIONS:
Drug: Induction chemotherapy - modified FOLFIRINOX regimen — An induction chemotherapy (6 cycles) combining irinotecan 180 mg/m2, oxaliplatin 85 mg/m2, elvorin 200 mg/m2 followed by a 46-hour continuous infusion 2,400 mg/m2) will be delivered every 15 days (D1=D15).
Other: Early tumor response evaluation by MRI volumetry — Two weeks after the CT completion, the tumor volume will be measured by MRI with specific software which automatically borders the tumor so as to determine the early tumor response. A centralized reassessment of all MRI exams will be systematically performed by two radiologists of the coordinator center.
Radiation: Radiochemotherapy Cap 50 — RCT Cap 50 will combine radiotherapy at a dose of 50 Gy by either conventional 3D or Intensity-Modulated RadioTherapy (IMRT) (2 Gy per fraction, 5 fractions per week during 5 weeks / 44 Gy in mini pelvis, and boost 6 Gy on reduced peritumoral volume) with concomitant oral capecitabine at 1600 mg/m2 per day delivered the days of radiotherapy treatment (2 daily intake).
  Arms: RCT Cap 50 and then rectal surgery
Procedure: Radical proctectomy with total mesorectal excision — The proctectomy can be performed by laparoscopic surgery or conventional laparotomy.

SUMMARY:
Locally advanced rectal carcinoma raise the issue of both the oncological control, local and general, and the therapeutic morbidity. Surgery alone can cure only one out of two patients, radiochemotherapy improves the local control but the metastatic risk remains about 30% with enhanced postoperative morbidity and poor functional results. The tumor response to preoperative treatment is the major prognostic factor which revealed the aggressiveness of the tumor. To this day, there are no biologic predictive markers for tumor response.

The purpose of this trial is to tailor the management according to the early tumoral response after short and intensive induction chemotherapy. MRI volumetric tumor response will be used to distinguish between good responders and bad responders.

"Very good" responders will be randomized to either immediate surgery or radiochemotherapy followed by surgery (Standard arm: Cap 50).

DETAILED DESCRIPTION:
Cancer of the rectum is a common disease. It affects nearly 15,000 new people each year, with more men (53%) than women (47%).

In more than 9 out of 10 cases, it occurs after 50 years. Three types of treatments are used to treat rectal cancer: surgery, radiotherapy and drug treatments.

The standard treatment for Locally Advanced Rectal Cancers (LARC) is multidisciplinary, combining chemotherapy, radiotherapy and surgery. The usual treatment in this situation is called induction chemotherapy administrated before radiochemotherapy. This phase of treatment taking place before surgery is called neoadjuvant therapy.

However, treating all cancers of the locally advanced rectum with the same neoadjuvant treatment exposes patients who are good responders to neoadjuvant chemotherapy with possible toxicity to radiotherapy and patients who are poor responders to ineffectiveness of conventional radiotherapy with surgery and so to a mutilating ineffective treatment.

The short- and long-term toxicity of pelvic radiation may be the most compelling reason to reconsider reflexive neoadjuvant radiochemotherapy (NA-RCT) and to move toward a more individualized approach.

A large North American trial is currently evaluating the suppression of preoperative radiation therapy in patients selected as a good responder to induction chemotherapy.

A first trial called GRECCAR-4 (Surgical Research Group on Rectum CAncer) with induction chemotherapy by 5 Fluorouracil + Irinotecan + Oxaliplatin and personalized radiochemotherapy reported the following results:

* High-dose induction chemotherapy is well tolerated and reproducible
* Early assessment after neo-adjuvant chemotherapy makes it possible to discriminate between good and bad responders without a negative impact on surgery.
* Personalized management of LARC according to the early tumor response to chemotherapy is possible.
* In good responder patients, a resection rate of 100% was achieved (even in the arm without radiotherapy), but due to poor recruitment, it is not possible to draw a formal conclusion regarding these promising results.
* The oncological results at 5 years show a local recurrence rate of 0% for the good responders and 4.8% for the poor responders. The 5-year overall survival was 86.7% with a 5-year progression-free survival of 75.0%.

GRECCAR 14 is the only French trial to question the feasibility of appropriate management of non-metastatic LARC. Its main objective is to evaluate, in good responder patients, personalized management after preoperative CT treatment.

GRECCAR-14 will try to confirm this strategy taking into account the 1st results of GRECCAR 4.

The study will initially focus on 200 patients to assess the surgical quality of this therapeutic strategy and then on 230 additional patients to assess the effectiveness of this personalized treatment on survival without recurrence.

ELIGIBILITY:
INCLUSION CRITERIA FOR SCREENING

1. Written consent,
2. Patient who receive Folfirinox,
3. Patient aged over 18 years old,
4. World Health Organization (WHO) performance status ≥ 1,
5. Histologically confirmed diagnosis of adenocarcinoma of the rectum,
6. Distal part of the tumor from 1 to 12 cm from the upper part of the levator ani (dynamic rectal examination),
7. No unequivocal evidence on CT-Scan of established metastatic disease,
8. MRI evaluation of the locally advanced tumor before neoadjuvant chemotherapy:

   1. Predictive CRM < 2 mm
   2. Or T3c-d (extending ≥ 5 mm beyond the muscularis propria) with extra mural venous invasion (EMVI)
   3. Or T4a-b (except bone and sphincteric invasion).

NON INCLUSION CRITERIA FOR SCREENING

1. Non measurable rectal tumor or not assessed by MRI before inclusion,
2. Ultra-low rectal tumor at diagnosis which imposes radiotherapy administration (inferior tumor pole less than 1 cm from the upper part of the levator ani).
3. Active cardiac disease including any of the following: a. Congestive heart failure ≥ New York Heart Association (NYHA) class 2 (appendix 4), b. Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months), c. Myocardial infarction less than 6 months before first dose of treatment, d. Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted),
4. Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 5 years prior to study inclusion, except for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non invasive tumor), Tis (carcinoma in situ) and T1 (lamina propria invasion)],
5. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months before start of treatment.

INCLUSION CRITERIA FOR EXPERIMENTAL TREATMENT

1. WHO performance status 0-1,
2. Patient with tumoral regression ≥ 60% and CRM ≥ 1mm,
3. No unequivocal evidence on CT-Scan of established metastatic disease,
4. General condition considered suitable for radical pelvic surgery and a systemic therapy with Capecitabine
5. Adequate hematologic, hepatic, renal and ionogram function assessed within 7 days prior to study treatment a. Platelet count ≥ 100,000/mm3; Hemoglobin (Hb) ≥ 9 g/dL; Absolute neutrophil count (ANC) ≥ 1,500/ mm3 b. Total bilirubin ≤ 1.5 x Upper Limit Normal (ULN), Alkaline phosphatases ≤ 3 x ULN and ASpartate aminoTransferase (AST) and ALanine aminoTransferase (ALT) ≤ 3 x ULN, c. Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance ≥ 50 ml/min according to Modification of Diet in Renal Disease (MDRD),
6. For women of reproductive potential, negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test obtained within 7 days before the start of study treatment. Women not of reproductive potential are female patients who are postmenopausal or permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy),
7. For women of childbearing potential and men, agreement to use an adequate contraception for the duration of study participation and up to 6 months following completion of therapy. Females of childbearing potential who are sexually active with a non-sterilized male partner must use 2 methods, of effective contraception. The investigator or a designated associate is requested to advise the patient on how to achieve an adequate birth control. Adequate contraception is defined in the study as any medically recommended method (or combination of methods) as per standard of care,
8. No evidence of chronic or acute ischemic heart disease,
9. Willing to participate to the study, and able to give informed consent and to comply with the treatment and follow-up schedules,
10. Affiliation to the French Social Security System.

NON-INCLUSION CRITERIA FOR EXPERIMENTAL TREATMENT

1. Patient with a history of pelvic radiotherapy,
2. Contraindication to chemotherapy and/or radiotherapy,
3. Complete or partial Dihydropyrimidine deshydrogenase (DPD) deficiency (uracilemia ≥ 16 ng/mL),
4. Any infection that could jeopardize treatment administration,
5. Any other serious concomitant disease or disorder that may interfere with the patient's participation in the study and safety during the study (e.g., severe liver, heart, kidney, lung, metabolic, or psychiatric disorders),
6. History of inflammatory bowel disease,
7. Patients with a history of pulmonary fibrosis or interstitial pneumonia,
8. Patients using antivitamin K (Coumadin etc…) but it's possible to substitute the antivitamin K treatment with low molecular weight heparins (LMWHs) before starting chemotherapy,
9. Known hypersensitivity to Capecitabine drug, study drug classes, or any constituent of the products,
10. Patient who received live attenuated vaccine within 10 days of inclusion,
11. Pregnant or breastfeeding woman. If a patient is of childbearing age, she must have a negative pregnancy test (serum β-hCG) documented 72 hours prior to inclusion,
12. Patient treated with an investigational drug within the last 30 days,
13. Patient under curatorship or guardianship or safeguard justice,
14. Inability to submit to medical monitoring of the trial for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1075 (Estimated)
Dates: Start 2021-11-26 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate (R0 is defined as Circumferential resection margin (CRM ≥ 1 mm) for Phase II | Within 15 days after surgery
  The excision limits will be determined precisely on the part, after exhaustive sampling of the maximum tumor extension zones and containing the surface of the inked mesorectum.
3-year Disease free survival (DFS) for Phase III | 3 years
  (DFS is defined as the time interval between randomization and the occurrence of the first event, such as local or metastatic recurrence, the development of a second cancer or death from any cause).Locoregional failure include locally progressive disease leading to an unresectable tumour, local R2 resection, or local recurrence after an R0-R1 resection.
  Patients without events at the time of analysis will be censored on the date of the last informative follow-up.

SECONDARY OUTCOMES:
Compliance rate with neoadjuvant treatment schedule | Within 4.5 months after the start of treatment
  To measure the compliance rate to the whole neoadjuvant schedule (induction CT + radiochemotherapy)
Pathological complete response rate | Within 15 days after surgery
  To assess the pathological complete response rate (ypT0N0)
Sphincter-saving surgery rate | Up to 2 months after the end of the neoadjuvant treatment
  To assess the impact of the therapeutic strategy on the rate of sphincter-saving surgery.
Quality of life by using the quality of life questionnaire score (QLQ-C30) | For a 1-year follow-up
  The EORTC QLQ-C30 uses for the questions 1 to 28 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome.
  The EORTC QLQ-C30 uses for the questions 29 and 30 a 7-points scale. The scale scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). Half points are not allowed. The range is 6. First of all, raw score has to be calculated with mean values. Afterwards linear transformation is performed to be comparable. More points are considered to have a better outcome.
Bowel function, Low anterior resection syndrome (LARS) | For a 1-year follow-up
  Assessed using LARS questionnaire (score 0-42, a high score indicates poor bowel function)
Quality of life by using the quality of life questionnaire score (QLQ-CR29) | For a 1-year follow-up
  Score 26-108, a high score indicates many symptoms of colorectal cancer.
3-year local recurrence free survival rate (L-RFS) | 3 years
  The time interval from the date of randomization to the date of local recurrence or death from any cause).Patients alive without local recurrence will be censored at the date of last follow-up.
3-year metastasis recurrence free survival rate (M-RFS) | 3 years
  The time interval from the date of randomization to the date of metastatic recurrence or death from any cause).Patients alive without metastasis will be censored at the date of last follow-up.
3-year Overall survival (OS) | 3 years
  The time interval from the date of randomization to the date of death from any cause. Patients alive will be censored at the date of last follow-up.
5-year Overall survival (OS) | 5 years
  The time interval from the date of randomization to the date of death from any cause. Patients alive will be censored at the date of last follow-up.
Local recurrence rate | For a 2-3-year follow-up
  The time interval from the date of randomization to the date of local recurrence. Patients without local recurrence will be censored at the date of last follow-up or death.
Clavien-Dindo grade | Within 1 month after surgery
  Grade 1 (light) to Grade 5 = Death of patient . It is widely used throughout surgery for grading adverse events (i.e. complications) which occur as a result of surgical procedures.
Neoadjuvant rectal Score by Fokas | Within 15 days after surgery
  The score uses the variables of clinical tumor stage, pathologic tumor stage, and pathologic nodal stage which are commonly available, furthering its utility in the clinical setting. The final scores range from 0 (good prognostic) to 100 (poor prognostic).
Rates of Total mesorectal excision (TME) grading according to Quirke | Within 15 days after surgery
  This grade is given by the pathologist on the appearance of the mesorectum on fresh specimen (complete grade = good resection), incomplete and near incomplete grade (between good and poor resection), incomplete grade = poor resection)
Distal margin to the tumor | Within 15 days after surgery
Definitive stoma rate | 36 MONTHS
Second surgery rate | 36 MONTHS
Rehospitalization rate | Within 1 month after surgery
Dworak Classification | Approximately 6 weeks after randomization
  Histopathologic analysis of tumor. Grade 0 to grade 4 with (Grade 4 = sterilized tumor to grade 0 = no regression of tumor)
Metastasis recurrence rate | For a 2-3-year follow-up
  the time to metastasis defined as the time interval from the date of randomization to the date of metastasis. Patients without metastasis will be censored at the date of last follow-up or death.
Disease Fee Survival rate (DFS) | For a 3-year follow-up
  the time interval from the date of randomization until the date of the first cancer-related event, or death from any cause). Patients alive without event will be censored at the date of last follow-up.
Assessment of adverse events by using the NCI-CTCAE version 5 scale | Approximately 72 months for all patients
  From the signature of informed consent until 60 days after Surgery
Evaluation of urinary function by International Prostate Symptom Score (IPSS) questionnaire score | For a 1-year follow-up
  Score 0-35, a high score indicates an impaired urinary function.
Evaluation of sexual function in men by International Index of Erectile Function (IIEFS) questionnaire score | For a 1-year follow-up
  Score 1-25, a low score indicates an impaired sexual function in men.
Evaluation of sexual function in women by Female Sexual Function Index (FSFI) questionnaire score | For a 1-year follow-up
  Score 4-95, a low score indicates an impaired sexual function in women.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Rouanet, MD, Study Chair — Philippe.Rouanet@icm.unicancer.fr
Locations (30):
- France (30):
  - Institut Paoli Calmettes, Marseille, Bouches Du Rhône
  - Hôpital Nord de Marseille, Marseille, Bouches Du Rhône
  - Hôpital Européen de MARSEILLE, Marseille, Bouches-du-rhône
  - CHU Besançon, Besançon, Doubs
  - CHU de Bordeaux, Bordeaux, Gironde
  - Insitut Régional du Cancer de Montpellier, Montpellier, Hérault
  - CHU de Nancy, Vandœuvre-lès-Nancy, Lorraine
  - Centre Alexis Vautrin, Nancy, Meurthe Et Moselle
  - Centre Oscart Lambret, Lille, Nord
  - CHU Amiens, Amiens, Picardie
  - CHU Clermont-Ferrand, Clermont-Ferrand, Puy De Dôme
  - CH PAU, Pau, Pyrénées-atlantiques
  - CHU de Lyon, Lyon, Rhône
  - CH Annecy, Annecy, Savoie
  - CHU Rouen, Rouen, Seine-Maritime
  - Hôpital Bicêtre, Le Kremlin-Bicêtre, Val De Marne
  - Bordeaux Colorectal Institute, Bordeaux
  - Centre Georges-François Leclerc, Dijon
  - Chu Grenoble, Grenoble
  - Chu Lille, Lille
  - CAC Léon Bérard, Lyon
  - Hôpital La Timone, Marseille
  - Centre Antoine Lacassagne, Nice
  - CHU de Nîmes, Nîmes
  - Hôpital Saint-Louis, Paris
  - Hôpital Saint-Antoine, Paris
  - Hôpital Européen Georges-Pompidou, Paris
  - Hôpital Diaconesses, Paris
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Yes
All data will be available after publication of the results in peer-reviewed revues, and in national and international meetings. It includes all disidentified participants' data, the study protocol, the statistical analysis plan and the analytic code. The corresponding author will provide data and datasets generated and/or analyzed during the study upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Access to study data upon written detailed request sent to ICM, following publication and until 5 years after publication of summary data.
Access Criteria: The data shared will be limited to that required for independent mandated verification of the published results, the applicant will need authorization from ICM for personal access, and data will only be transferred after signing of a data access agreement.

REFERENCES:
- [Background] Sauer R, Liersch T, Merkel S, Fietkau R, Hohenberger W, Hess C, Becker H, Raab HR, Villanueva MT, Witzigmann H, Wittekind C, Beissbarth T, Rodel C. Preoperative versus postoperative chemoradiotherapy for locally advanced rectal cancer: results of the German CAO/ARO/AIO-94 randomized phase III trial after a median follow-up of 11 years. J Clin Oncol. 2012 Jun 1;30(16):1926-33. doi: 10.1200/JCO.2011.40.1836. Epub 2012 Apr 23. PMID 22529255
- [Background] Rodel C, Graeven U, Fietkau R, Hohenberger W, Hothorn T, Arnold D, Hofheinz RD, Ghadimi M, Wolff HA, Lang-Welzenbach M, Raab HR, Wittekind C, Strobel P, Staib L, Wilhelm M, Grabenbauer GG, Hoffmanns H, Lindemann F, Schlenska-Lange A, Folprecht G, Sauer R, Liersch T; German Rectal Cancer Study Group. Oxaliplatin added to fluorouracil-based preoperative chemoradiotherapy and postoperative chemotherapy of locally advanced rectal cancer (the German CAO/ARO/AIO-04 study): final results of the multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2015 Aug;16(8):979-89. doi: 10.1016/S1470-2045(15)00159-X. Epub 2015 Jul 15. PMID 26189067
- [Background] Martin ST, Heneghan HM, Winter DC. Systematic review and meta-analysis of outcomes following pathological complete response to neoadjuvant chemoradiotherapy for rectal cancer. Br J Surg. 2012 Jul;99(7):918-28. doi: 10.1002/bjs.8702. Epub 2012 Feb 23. PMID 22362002
- [Background] Bregendahl S, Emmertsen KJ, Lous J, Laurberg S. Bowel dysfunction after low anterior resection with and without neoadjuvant therapy for rectal cancer: a population-based cross-sectional study. Colorectal Dis. 2013 Sep;15(9):1130-9. doi: 10.1111/codi.12244. PMID 23581977
- [Background] Chen TY, Wiltink LM, Nout RA, Meershoek-Klein Kranenbarg E, Laurberg S, Marijnen CA, van de Velde CJ. Bowel function 14 years after preoperative short-course radiotherapy and total mesorectal excision for rectal cancer: report of a multicenter randomized trial. Clin Colorectal Cancer. 2015 Jun;14(2):106-14. doi: 10.1016/j.clcc.2014.12.007. Epub 2014 Dec 31. PMID 25677122
- [Background] Schrag D, Weiser MR, Goodman KA, Gonen M, Hollywood E, Cercek A, Reidy-Lagunes DL, Gollub MJ, Shia J, Guillem JG, Temple LK, Paty PB, Saltz LB. Neoadjuvant chemotherapy without routine use of radiation therapy for patients with locally advanced rectal cancer: a pilot trial. J Clin Oncol. 2014 Feb 20;32(6):513-8. doi: 10.1200/JCO.2013.51.7904. Epub 2014 Jan 13. PMID 24419115
- [Background] Weiser MR, Fichera A, Schrag D, Boughey JC, You YN. Progress in the PROSPECT trial: precision treatment for rectal cancer? Bull Am Coll Surg. 2015 Apr;100(4):51-2. No abstract available. PMID 25939207
- [Background] Rouanet P, Rullier E, Lelong B, Maingon P, Tuech JJ, Pezet D, Castan F, Nougaret S; and the GRECCAR Study Group. Tailored Treatment Strategy for Locally Advanced Rectal Carcinoma Based on the Tumor Response to Induction Chemotherapy: Preliminary Results of the French Phase II Multicenter GRECCAR4 Trial. Dis Colon Rectum. 2017 Jul;60(7):653-663. doi: 10.1097/DCR.0000000000000849. PMID 28594714
- [Background] Kang JH, Kim YC, Kim H, Kim YW, Hur H, Kim JS, Min BS, Kim H, Lim JS, Seong J, Keum KC, Kim NK. Tumor volume changes assessed by three-dimensional magnetic resonance volumetry in rectal cancer patients after preoperative chemoradiation: the impact of the volume reduction ratio on the prediction of pathologic complete response. Int J Radiat Oncol Biol Phys. 2010 Mar 15;76(4):1018-25. doi: 10.1016/j.ijrobp.2009.03.066. Epub 2009 Aug 3. PMID 19647949
- [Background] Rouanet P. Which Trial to Demonstrate the Truthfulness of a Tailored Strategy in Rectal Carcinoma? Dis Colon Rectum. 2018 Jan;61(1):e1-e2. doi: 10.1097/DCR.0000000000000977. No abstract available. PMID 29219925
- [Background] Nougaret S, Castan F, de Forges H, Vargas HA, Gallix B, Gourgou S, Rouanet P; GRECCAR Study Group. Early MRI predictors of disease-free survival in locally advanced rectal cancer from the GRECCAR 4 trial. Br J Surg. 2019 Oct;106(11):1530-1541. doi: 10.1002/bjs.11233. Epub 2019 Aug 22. PMID 31436325
- [Background] Fokas E, Glynne-Jones R, Appelt A, Beets-Tan R, Beets G, Haustermans K, Marijnen C, Minsky BD, Ludmir E, Quirke P, Sebag-Montefiore D, Garcia-Aguilar J, Gambacorta MA, Valentini V, Buyse M, Rodel C. Outcome measures in multimodal rectal cancer trials. Lancet Oncol. 2020 May;21(5):e252-e264. doi: 10.1016/S1470-2045(20)30024-3. PMID 32359501
- [Background] Rouanet P, Castan F, Mazard T, Lemanski C, Nougaret S, Deshayes E, Chalbos P, Gourgou S, Taoum C; GRECCAR, PRODIGE study group. GRECCAR 14 - a multicentric, randomized, phase II-III study evaluating the tailored management of locally advanced rectal carcinoma after a favourable response to induction chemotherapy: Study protocol. Colorectal Dis. 2023 Oct;25(10):2078-2086. doi: 10.1111/codi.16740. Epub 2023 Sep 11. PMID 37697712